CLINICAL TRIAL: NCT06558864
Title: The Efficacy and Safety of Subiculum Stereotactic-EEG Guided Radio-frequency Thermocoagulation for Mesial Temporal Lobe Epilepsy With Hippocampus Sclerosis: A Prospective, Single-Arm Trial
Brief Title: High Selective Subiculum SEEG Guided RF-TC for mTLE-HS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-174-002
Record Dates: First submitted 2024-08-04; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-07

CONDITIONS: Mesial Temporal Lobe Epilepsy With Hippocampal Sclerosis; Epilepsy
Keywords: Radio-frequency thermocoagulation; Stereoelectroencephalography; Subiculum
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subiculum RF-TC group (Experimental): SEEG recording and Subiculum RF-TC minimal invasive treatment for mTLE-HS
  Interventions: Procedure: Subiculum RF-TC

INTERVENTIONS:
Procedure: Subiculum RF-TC — SEEG implantation after evaluation, record the interictal and ictal EEG, and perform Subiculum RF-TC.

SUMMARY:
The primary objective of this research is to study the efficacy and safety of Stereotactic EEG (SEEG) guided radio-frequency thermocoagulation (RF-TC) of Subiculum as adjunctive therapy for reducing the frequency of seizures in drug-resistant temporal lobe epilepsy with Mesial temporal lobe epilepsy with hippocampal sclerosis (mTLE-HS).

DETAILED DESCRIPTION:
Mesial temporal lobe epilepsy (mTLE) is the most classical subtype of temporal lobe epilepsy, which is the indication of surgical intervention after evaluation. This project aims to include 20 participants, and evaluate the effectiveness and safety of Stereotactic EEG (SEEG) guided radio-frequency thermocoagulation (RF-TC) of Subiculum in patients with mesial temporal lobe epilepsy with hippocampal sclerosis through A prospective, interventional, unblinded, single-arm clinical trial. It is expected to provide new therapeutic options for patients with mTLE-HS with alternative treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Participants are between the ages of 14 -65 years of age
* Refractory to anti-seizure medications (ASMs).
* Persistence of disabling seizures at least 2 times per month during the Baseline Phase，with no more than 30 days between seizures during the Baseline Phase.
* Hippocampal atrophy on MRI T1 imaging with increased ipsilateral mesial signal on T2 imaging
* Interictal EEG shows focal or lateralized spikes on temporal, frontal zone, or sphenoid electrode
* Ictal EEG onset is focal or lateralized on the ipsilateral side
* Ipsilateral temporal focal hypometabolism on PET
* Must be agreed by a consensus of ipsilateral mesial temporal origin by a multidisciplinary discussion

Exclusion Criteria:

* Diagnosed with generalized or hereditary epilepsy with ion channel gene mutations;
* Psychogenic non-epileptic seizures within 12 months;
* Presence of implanted electrical stimulation medical device anywhere in the body (e.g., pacemaker, spinal cord stimulator, responsive neurostimulation) or any metallic implants in the head (e.g., aneurysm clips, cochlear implants). Note: Vagal nerve stimulators are allowed if the parameter remains stable for at least 3 months prior to the screening visit;
* Risk factors that would put the participant at risk for intraoperative or postoperative bleeding. (e.g., coagulation abnormalities, etc.) or the need for chronic anticoagulation or antiplatelet aggregation medications;
* IQ < 55 or severe cognitive dysfunction, unable to complete the study;
* Diagnosed with a progressive neurological disorder (including progressive Rasmussen's encephalitis, etc.);
* Diagnosed with a severe neuropsychiatric disorder such as dementia, major depression (admission to a psychiatric specialty/hospital within 5 years or any suicidal or self-injurious tendencies), schizophrenia, or neurodegenerative disorders;
* Diagnosed with other serious physical disorders, internal diseases or severe abnormalities in liver or kidney function;
* Pregnant, or planning to pregnant within 2 years;
* Participation in another clinical study within 3 months;
* Not suitable for enrollment as assessed by the multidisciplinary team of the center.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-09 (Estimated); Primary Completion 2025-08-20 (Estimated); Study Completion 2027-08-20 (Estimated)

PRIMARY OUTCOMES:
Seizure frequency (SF28) | Up to 1 year after subculum-SEEG Guided RF-TC
  Seizure frequency (SF28) is defined as seizure count per month (28-day) period. The SF28 is calculated as follows, where D=total number of days for which seizure information is collected for the specific 28-day interval:
  SF28=(Total number of seizures in D days/D)*28. In addition, the baseline seizure frequency is defined as mean of 3-month SF28 in the baseline period. The seizure frequency in double-blind phase is defined as SF28 per month during the double-blind period. Percent change in seizure frequency=100*(double-blind SF28-baseline SF28)/baseline SF28.

SECONDARY OUTCOMES:
Seizure Responder Rate | Up to 1 year after subculum-SEEG Guided RF-TC
  The proportion of patients with a ≥ 50% reduction from Baseline in seizure frequency.
Life quality evaluation | Up to 1 year after subculum-SEEG Guided RF-TC
  Percentage change from baseline in Quality of Life in Epilepsy-31 inventory (QOLIE-31) score.
Cognitive function evaluation (MMSE) | Up to 1 year after subculum-SEEG Guided RF-TC
  Percentage change from baseline in Mini-Mental State Examination (MMSE) score.
Cognitive function evaluation (MoCA) | Up to 1 year after subculum-SEEG Guided RF-TC
  Percentage change from baseline in Montreal Cognitive Assessment (MoCA) score.
Adverse Events | Up to 1 year after subculum-SEEG Guided RF-TC
  Rate of adverse events which were judged to be study-related throughout the study.
Incidence of Sudden Unexpected Death in Epilepsy (SUDEP) | Up to 1 year after subculum-SEEG Guided RF-TC
  The number presented is for Definite and Probable SUDEP. The rate is calculated per 1000 subject years of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Liankun Ren, MD, Principal Investigator — Xuanwu Hospital, Beijing